CLINICAL TRIAL: NCT01215825
Title: The Therapeutic Impact of Various Doses of Systemic Steroid in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: The Doses of Systemic Steroid in Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD)
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Ping-huai Wang, Far Eastern Memorial Hospital
Other Study IDs: 098097-3
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; systemic steroid
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HD, LD, NIL: HD: the highest daily dose of steroids receiving more than 60 mg/day LD: the highest daily dose of steroids receiving less or equal to 60 mg/day NIL: no steroid use

SUMMARY:
It is well established that steroid use is a benefit in the treatment of chronic obstructive pulmonary disease (COPD) with acute exacerbation (AE). But it is still debated about the regimen and dosage of steroid use. From this retrospective review of medical charts, the researchers investigated the therapeutic impact of various steroid dosages in COPD with AE.

DETAILED DESCRIPTION:
Data collection from medical charts was conducted at Far Eastern Memorial Hospital, a tertiary-care hospital with around 900 beds. Patients who were admitted from January 2008 to December 2008 and diagnosed as having chronic obstructive pulmonary disease with acute exacerbation (code ICD-9: 491.21) were included in this study. The study was approved by the Institutional Review Board of the Far Eastern Memorial Hospital (FEMH:098097-3).

Demographic data, medical histories and medicine prescriptions at outpatient clinics, emergency and inpatient departments were collected. The initial presentations of acute exacerbation and laboratory data were also summarized from the records of the emergency department. The reports of pulmonary function tests within 6 months before or after the exacerbations were included while reviewing the charts. The probability of concomitant pneumonia (pAECOPD) was determined by attending physicians and reviewed by the investigator according to the radiologic findings. If there were incoherent opinions about the probability of pneumonia between the physicians and the investigator, it was determined by another independent pulmonologist. The highest daily doses and total doses of systemic steroids were calculated and recorded as the equivalent doses of prednisolone (1 mg methylprednisolone is equal to 1.25 mg prednisolone; 1 mg hydrocortisone is equal to 0.25 mg prednisolone). The subjects were divided into 3 groups according to the highest daily dose of steroids as follows: patients receiving more than 60 mg/day were designated to the HD group; those receiving less than or equal to 60 mg/day to the LD group; and those who did not receive any steroids during admission to the NIL group. The length of stay (LOS) was defined as the duration from admission to the emergency department to discharge. Hyperglycemia, psychosis, nosocomial infections and active peptic ulcer diseases were regarded as acute side effects of systemic steroids. Hyperglycemia was defined as a new blood sugar level of more than 200 mg/dl in patients without a history of diabetic mellitus, or an increment in diabetes medications. The relapse rate within 30 days was assessed by outpatient follow-up records.

ELIGIBILITY:
Inclusion Criteria:

* From January 2008 to December 2008, patients were admitted and diagnosed as having chronic obstructive pulmonary disease with acute exacerbation (code ICD-9: 491.21)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2008 to December 2008, patients were admitted and diagnosed as having chronic obstructive pulmonary disease with acute exacerbation (code ICD-9: 491.21)
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

SECONDARY OUTCOMES:
side effects | 2009
  the side effects of the systemic steroids within groups with different steroid regimens.
30-day relapse rates | 2009
  the 30-day relapse rates within groups of various steroid doses

CONTACTS AND LOCATIONS:
Overall Officials: Ping-huai Wang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Ban-chiao City, Taipei, Taiwan